CLINICAL TRIAL: NCT07006311
Title: Robotic-assisted Bronchoscopy Under Moderate Sedation With Propofol: A Single-center Pilot Study.
Brief Title: Robotic-assisted Bronchoscopy Under Moderate Sedation With Propofol
Acronym: Robofol
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: BASEC-Nr: 2025-D0013
Record Dates: First submitted 2025-05-14; First posted 2025-06-05 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Lung Lesions; Robotic Assisted Bronchoscopy; Propofol; Bronchoscopy; Bronchoscopy Biopsy
Keywords: Robotic-assisted bronchoscopy; robotic assisted bronchoscopy; diagnosis of lung lesions; moderate sedation

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Robotic-assisted bronchoscopy with Propofol (Experimental)
  Interventions: Device: Robotic-assisted bronchoscopy under propofol

INTERVENTIONS:
Device: Robotic-assisted bronchoscopy under propofol — In this study, patients will undergo a robotic-assisted bronchoscopy under moderate sedation with propofol. While the use of propofol as a sedative is common for manual bronchoscopies, robotic-assisted bronchoscopy is only permitted under general anesthesia. In the study intervention, the investigators want to test the feasibility of the combination of robotic-assisted bronchoscopy under propofol.

SUMMARY:
In this study, the investigators want to find out whether robot-assisted bronchoscopy also works with moderate sedation (Propofol), as is already used in standard bronchoscopies. The study is being conducted as a pilot study. This means that it is an initial test run for a scientific investigation. The investigators are testing on a small scale whether the intervention works as predicted before a larger study is conducted.

ELIGIBILITY:
Inclusion Criteria:

* informed consent signed by the subject
* aged at least 18 years
* scheduled for bronchoscopy with moderate sedation and tracheal intubation in order to obtain at least 1 specimens of the lung via transbronchial biopsy
* necessary periinterventional laboratory examinations needed for the bronchoscopy
* judgement of the subject

Exclusion Criteria:

* endobronchial lesion causing lobar atelectasis
* inability or contraindications to undergo bronchoscopy (e.g. severe cardiopulmonary diseases, coagulation disorders, intolerance to anesthesia or endoscopic operation, psychiatric disorders or severe neurosis)
* pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-14 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Confirmation of tool-in-lesion | during the intervention
  Composite outcome defined as meeting at least one of the following criteria: 1) Radiological confirmation of the biopsy tool located within the target lung lesion using cone-beam CT. 2) Positive signal on radial endobronchial ultrasound (rEBUS) indicating the lesion was reached. 3) Pathological confirmation of specific malignant or benign tissue in the biopsy sample.
Acquisition of at least one histological sample | during the intervention
histopathological classification of the pulmonary lesion | From enrollment to the end of treatment at 8 days.

SECONDARY OUTCOMES:
Procedure duration | during the intervention
Diagnostic yield of biopsies | From enrollment to the end of treatment at 8 days.
  According to the ATS2024 strict consensus criteria (https://doi.org/10.1164/rccm.202401-0192ST)
diagnostic accuracy for malignancy | From enrollment to the end of treatment of 3 months
  Biopsies with definitive malignancy/Cases with proven malignance over the course of 3 months
cost analysis | From enrollment to the end of treatment at 8 days.
  Total billed costs in CHF for the bronchoscopy excl. anesthesia
Safety profile | From enrollment to the end of treatment at 8 days.
  Rate of pneumothoraces, bleeding rates (Nashville Classification Grad >2), and rate of unplanned hospitalizations >5 days.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland